CLINICAL TRIAL: NCT01080053
Title: Observational Study to Determine the Relationship Between the Degree of Disability and the Presence of Sexual Dysfunction and Between Sexual Dysfunction and the Quality of Life in Patients With Multiple Sclerosis (RRMS)
Brief Title: Sexual Dysfunction, Disability and Quality of Life in Patients With Multiple Sclerosis (MS)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Quimica Argentina S.A.I.C (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200077-511
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis, Relapsing Remitting
Keywords: Multiple Sclerosis, Relapsing Remitting; Sexual dysfunction
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is an observational, prospective, non-interventional, non-controlled study planned to be conducted in subjects with Relapsing-Remitting Multiple Sclerosis (RRMS).

The purpose of this observational study is to determine the correlation between the degree of disability and sexual dysfunction; and between the sexual dysfunction and the quality of life (QoL) of subjects with Relapsing Remitting Multiple Sclerosis (RRMS) in Argentina.

DETAILED DESCRIPTION:
Multiple sclerosis, like most of the chronic diseases, can affect the sexuality of those who suffer from it. This situation has an evident and marked impact on the QoL of the subjects and his/her partner, and causes conflict in the relationship, with high levels of mutual dissatisfaction.

The impact that the duration of the disease or the degree of disability have on the level of sexual dysfunction is not clear. However, the possible organic and state of mind causes of the sexual dysfunction makes us think that the degree of disability is a crucial factor in the genesis and duration of the symptoms in the sexual area. The frequency with which the sexual dysfunction is detected or referred in these subjects is variable.

The sexual dysfunction in subjects with MS is typically characterized by a decreased libido, erectile dysfunction and ejaculation disorders in men, and decreased lubrication and anorgasmia in women. The most commonly detected problems are the erectile dysfunction and/or lack of sexual interest in men and lack of interest, decreased libido and orgasmic disorder in women.

This observational study aims to assess a population of subjects with MS that show symptoms of sexual dysfunction, in order to determine the relationship, if any, between the severity of the general disability and the incidence of sexual dysfunction. At the same time, this epidemiologic study aims to measure the impact the sexual dysfunction generates in the quality of life of subjects with MS.

The data to be obtained could contribute to a better understanding of the relationship between the studied variables and, eventually, to alert the treating doctors about the incidence of these morbid associations.

The total duration of the study is 24 months. The recruiting period will be 12 months. Once the recruiting time is over, the collection of data will continue during the full 24 months period that was planned.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 21 years of age
* Subjects with established diagnosis of RRMS according to the revised McDonald criteria - 2005
* Subjects with a diagnosis of RRMS for more than one year
* The subject who have signed the Informed Consent

Exclusion Criteria:

* Subjects with no sexual experience
* Subjects with other diseases associated to MS
* Subjects with psychiatric diseases that could cause sexual dysfunction
* Subjects with one relapse during the previous month
* Use of antidepressants and/or corticosteroids during the previous month

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with established diagnosis of RRSM for more than one year.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2008-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The correlation between the degree of disability and sexual dysfunction, and between the sexual dysfunction and the QoL of subjects | Initial visit (Day 0) and each follow up visit upto the observation period of 24 months
  Mini-Mental State Examination (MMSE) Psychotropic-Related Sexual Dysfunction Questionnaire (PRSexDQ) Hamilton Rating Scale for Depression (HRSD)

CONTACTS AND LOCATIONS:
Overall Officials: Norma Deri, PhD, Principal Investigator
Locations (1):
- Dr. Norma Deri, Buenos Aires, Argentina